CLINICAL TRIAL: NCT05590143
Title: Preoperative Sodium Glucose Cotransporter 2 Inhibitors for Prevention of Postoperative Acute Kidney Injury in Cardiac Surgery Patients - a Randomized, Placebo-controlled, Multi-centre, Phase IV Clinical Trial
Brief Title: proMoting Effective Renoprotection in Cardiac sURgery Patients by Inhibition of SGLT-2
Acronym: MERCURI-2
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Abraham Hulst, MD, PhD, Principal Investigator, Amsterdam UMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MERCURI-2; 2022-002453-25 (EudraCT Number); 2024-515260-31-00 (EU CTIS Number); 10140022010003 (Other Grant/Funding Number: Netherlands Organisation for Health Research and Development); NL81190.018.22 (Registry Identifier: Central Committee on Research Involving Human Subjects); 2022.0795 (Other: Medical Ethics Committee Amsterdam UMC)
Record Dates: First submitted 2022-10-10; First posted 2022-10-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Cardiac Surgery; Sodium-Glucose Transporter 2 Inhibitor
Keywords: Cardiac Surgery; Acute Kidney Injury; SGLT2i; Dapagliflozin
MeSH Terms: conditions — Acute Kidney Injury | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga]
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga] — One oral tablet, once daily starting one day prior to surgery and continued until two days postoperatively (four doses).
  Other Names: Farxiga; SGLT2i; Sodium glucose co-transporter-2 inhibitor
  Arms: Intervention
Drug: Placebo — One oral tablet, once daily starting one day prior to surgery and continued until two days postoperatively (four doses).
  Arms: Placebo

SUMMARY:
Multi-centre, triple-blinded (patients, physicians, investigators), parallel-group, balanced (1:1), stratified (sex, type 2 diabetes mellitus), randomized, controlled (placebo), phase IV clinical trial to investigate the potential of preoperative initiation (from day 1 before surgery) and perioperative continuation (until day 2 after surgery) of the SGLT2 inhibitor dapagliflozin 10 mg once daily to prevent AKI according to the KDIGO criteria (an increase in serum creatinine by 0.3 mg/dl (26.5 mmol/l) within 48 hours; or an increase in serum creatinine to 1.5 times baseline, within 7 days; or a urine output <0.5 ml/kg/h for >6 hours) in adult (>18 years old) patients undergoing cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
Background of the study:

Acute kidney injury is one of the most common complications after cardiac surgery. The new glucose-lowering therapy, sodium glucose transport protein 2 inhibitors (SGLT2i) possess renoprotective properties in people with chronic kidney disease in the presence or absence of type 2 diabetes. Large cardiovascular outcome trials in patients with diabetes observed a lower incidence of acute kidney injury. However, these studies were not powered to investigate this nor did acute kidney injury concern an adjudicated endpoint.

Objective of the study:

To investigate the potential of preoperative initiation (from day 1 before surgery) and perioperative continuation (until day 2 after surgery) of the SGLT2 inhibitor dapagliflozin 10 mg once daily to prevent AKI according to the KDIGO criteria in patients undergoing cardiopulmonary bypass surgery.

Study design:

Multi-centre, triple-blinded (patients, physicians, investigators), parallel-group, balanced (1:1), stratified (sex, type 2 diabetes mellitus), randomized, controlled (placebo), phase IV clinical trial.

Study population:

Patients undergoing cardiac surgery, aged >18 years-old.

Intervention:

Participants receive 10 mg dapagliflozin once daily or matching placebo starting 1 day prior to surgery and continued until two days postoperatively (four doses).

Primary outcome of the study:

Incidence of AKI occurring in 7 days after surgery, according to KDIGO criteria, defined as an increase in serum creatinine by 0.3 mg/dl (26.5 mmol/l) within 48 hours; or an increase in serum creatinine to 1.5 times baseline, within 7 days; or a urine output <0.5 ml/kg/h for >6 hours.

Secondary outcomes of the study:

1. Incidence of Stage 3 AKI.
2. Postoperative change of eGFR.
3. Postoperative Atrial Fibrillation for which treatment is initiated.
4. Length of Stay in the Intensive Care Unit.
5. Length of Stay in hospital.
6. MAKE: Major Adverse Kidney Events
7. MACE: Major Adverse Cardiovascular Events
8. Patient-reported quality of recovery 1: DAH30: Days at Home in first 30 days
9. Patient-reported quality of recovery 2: WHO-DAS 2.0: World Health Organisation Disability Assessment Schedule 2.0
10. Patient-reported quality of recovery 3: EQ5D5L: 5 level EuroQol 5D questionnaire.
11. Safety outcomes: incidence of genital mycotic infections, diabetic keto-acidosis, hypoglycaemia, postoperative complications and Serious Adverse Events (SAEs).
12. Productivity costs
13. Healthcare costs
14. Hyperglycaemia (> 10 mmol/l)
15. Hypoglycaemia (< 4 mmol/l)
16. Heart Rate
17. Mean Arterial Pressure
18. Cardiac Output
19. Peak postoperative Troponin
20. Peak postoperative CK-MB
21. Postoperative Left Ventricular Function
22. Urinary oxygenation (patients included at Amsterdam UMC only)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

General trial-related burden:

The investigators will withdraw 4.5 mL of blood at one day before surgery and one day postoperatively for biomarker analysis. No extra venepunctures are required, as these measurements coincide with routine clinical care.

Intervention group-related burden:

Participants will be asked to take either 1 tablet of 10 mg dapagliflozin once daily from 1 days before surgery until 2 days postoperative (including the day of surgery, four doses total) or a matching placebo regimen. Patients randomized to dapagliflozin will run a small risk of treatable side effects related to the study drug. These are rare for short-term treatments. Participants will be informed about the following side effects:

1. Genital mycotic infections: these usually only occur after longer-term use of SGLT2 inhibitors. In this study, patients will only receive this medication for up to 10 doses. Treatment of this side effect is straightforward with antifungal treatment.
2. Euglycemic ketoacidosis: a lowering of the pH in the blood through the build-up of ketones. This has been described in patients on long-term treatment and is ascribed to altered insulin sensitivity through increased glucose loss by SGLT2 inhibition. For this and other reasons, patients with type 1 diabetes mellitus and patients with type 2 diabetes mellitus and a body mass index <25 kg/m2 are excluded from this trial. We will monitor perioperative glucose and pH levels in all participants according to routine perioperative care. In addition, patients using insulin therapy will receive a perioperative glucose/insulin infusion, which suppresses ketone production. Should keto acidosis occur in any other patient, treatment is straightforward with a glucose-insulin infusion.
3. Hypoglycemia: only patients with diabetes mellitus using sulfonylurea or insulin are at risk, according to previous research. To prevent this side effect: patients will receive an individualized adaptation of their glucose-lowering medication by the investigator team. To treat this side effect, blood glucose will be monitored in all patients according to standard perioperative cardiac surgery care and hypoglycaemia treatment protocols with urgent administration of intravenous glucose are in place.

Risk-benefit:

There is solid evidence to support that SGLT2 inhibitors offer kidney protection. Acute kidney injury is a common complication after cardiac surgery. The investigator's hypothesis is, therefore, that patients in the intervention group will receive protection against acute kidney injury. In addition, the results from this trial could lead to the improvement of care and protection of future patients undergoing cardiac surgery. The side-effect profile of dapagliflozin is mild, and participants will be intensively monitored in this study. Therefore, the investigators estimate that the benefits outweigh the risks of participation in this trial.

Relevance and intended applications:

The aim of this study is to determine whether SGLT2i can reduce the incidence of AKI following cardiac surgery. Based on the results of this trial, SGLT2 inhibitors can be applied as a standard prophylactic treatment in cardiac surgery patients to prevent AKI.

Sample size:

The investigators expect an incidence of AKI in the placebo group of 22%, as a conservative estimation, based on previous cohorts. Large outcome trails found a relative risk reduction for AKI of 0.64 with SGLT2 inhibition. This translates into an absolute risk reduction of 7.9% and an expected incidence in the intervention group of 14.1%. The required total sample size to find such a difference based on Fisher Exact test, with two-sided alpha at 0.05 and 80% power is 784. Therefore, the aim is to include 392 patients per arm.

Keywords: SGLT2i; Acute Kidney Injury (AKI); Cardiac Surgery

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years-old
2. Undergoing elective cardiac surgery.
3. Providing informed consent

Exclusion Criteria:

1. Current treatment with SGLT2 inhibitors
2. Reduced kidney function at baseline with eGFR < 20 ml/min at time of inclusion
3. Diabetes Mellitus Type 1
4. History of diabetic keto acidosis
5. Diabetes Mellitus Type 2 with BMI<25 for people with type 2 diabetes who are using multiple daily insulin injections (both short and long-acting insulin)
6. Systolic blood pressure < 100 mmHg at time of inclusion
7. Emergency surgery, defined as in need of surgery for medical reasons < 7 days, i.e. "S1-4" according to the Amsterdam UMC classification
8. Female of child-bearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
9. Known or suspected allergy to trial products or other drugs in the same class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
AKI | Recorded daily until day 7 postoperatively or until discharge from hospital (earlier).
  Incidence of Acute Kidney Injury (AKI) occurring in 7 days after surgery, according to KDIGO criteria, defined as an increase in serum creatinine by 0.3 mg/dl (26.5 mmol/l) within 48 hours; or an increase in serum creatinine to 1.5 times baseline, within 7 days; or a urine output <0.5 ml/kg/h for >6 hours.

SECONDARY OUTCOMES:
AKI-3 | Recorded daily until day 7 postoperatively or until discharge from hospital (earlier).
  Incidence of Stage 3 AKI according to KDIGO (Kidney Disease Improving Globel Outcomes) criteria.
eGFR | Recorded daily until day 7 postoperatively or until discharge from hospital (earlier).
  Postoperative maximum change of estimated Glomerular Filtration Rate (eGFR) compared to the baseline eGFR.
AF | Recorded daily until day 7 postoperatively or until discharge from hospital (earlier).
  Postoperative Atrial Fibrillation (AF) defined as any episode for which treatment is initiated.
LoS-ICU | Recorded on day of discharge from ICU, assessed up to 30 days.
  Length of Stay in the Intensive Care Unit (LoS-ICU), measured in days from transfer to ICU.
LoS-Hos | Recorded on day of discharge from the hospital, assessed up to 30 days.
  Length of Stay in the Hospital, measured in days from admission to hospital.
MAKE | Within 30 days postoperatively.
  Major Adverse Kidney Events (MAKE). Composite endpoint of death, new dialysis, and worsened renal function.
MACE | Within 30 days postoperatively.
  Major Adverse Cardiovascular Events (MACE). Composite endpoint of cardiovascular death, nonfatal myocardial infarction (MI), nonfatal ischaemic cerebral vascular accident (iCVA) and hospitalization for heart failure.
QoR 1: DAH30 | Recorded at 30 days postoperatively.
  Patient-reported quality of recovery, according DAH30: Days at Home in first 30 days.
QoR 2: WHODAS2 | Recorded at 30 days postoperatively.
  Patient-reported Quality of Recovery (QoR), according to World Health Organisation Disability Assessment Schedule 2.0 (WHO-DAS2.0). Summarized in a score between 0 - 100 with 0 being the best score (no disability) and 100 the worst (maximal disability).
QoR 3: EQ5D5L | Recorded at 30 days postoperatively.
  Patient-reported Quality of Recovery (QoR), according to 5 level EuroQol 5D questionnaire (EQ5D5L): a standardised measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. Summarized in a score between 0 - 1 with 0 being the best score (no disability) and 1 the worst (maximal disability).
Safety outcomes | Within 30 days postoperatively.
  Genital mycotic infections, diabetic keto-acidosis, and hypoglycaemia, in addition to incidence of postoperative complications and Serious Adverse Events (SAEs)
Health care costs | Recorded at 30 days postoperatively.
  Healthcare costs will be objectified to weigh cost-effectiveness, using the iMCQ:
  * IMCQ: IMTA (Institute for Medical Technology Assessment) Medical Consumption Questionnaire
Productivity costs | Recorded at 30 days postoperatively.
  Productivity costs will be objectified to weigh cost-effectiveness, using the iPCQ: IMTA (Institute for Medical Technology Assessment) Productivity Cost Questionnaire
Hypoglyceamia | From admission to hospital until day 3 postoperatively.
  Incidence of hypoglycaemia (blood glucose < 4 mmol/l) detected during routine peri-operative glucose measurements.
Hyperglyceamia | From admission to hospital until day 3 postoperatively.
  Incidence of hyperglycaemia (blood glucose > 10 mmol/l) detected during routine peri-operative glucose measurements.
Haemodynamics 1: HR | From start of anaesthesia until discharge from the Intensive Care Unit, assessed up to 72 hours.
  Peri-operative hourly average heart rate (HR, beats per minute) from the start of anaesthesia until discharge from the Intensive Care Unit.
Haemodynamics 2: MAP | From start of anaesthesia until discharge from the Intensive Care Unit, assessed up to 72 hours.
  Peri-operative hourly average mean arterial blood pressure (MAP, mmHg) from start of anaesthesia until discharge from the Intensive Care Unit.
Haemodynamics 3: CO | From start of anaesthesia until discharge from the Intensive Care Unit, assessed up to 72 hours.
  Peri-operative average hourly cardiac output (CO, l/min) from start of anaesthesia until discharge from the Intensive Care Unit.
Cardiac biomarker 1: Troponin | From transfer to ICU until 48 hours postoperatively.
  Peak troponin concentration, routinely measured during clinical practice.
Cardiac biomarker 2: CK-MB | From transfer to ICU until 48 hours postoperatively.
  Peak CK-MB concentration, as routinely measured during clinical practice.
Postoperative LVF | Within 30 days postoperatively.
  Qualitative assessment (categorised as normal, or mildly, moderately or severely reduced function) of left ventricular function (LVF) as noted by the echocardiographer for routinely performed postoperative echocardiography performed during routine follow-up.
Urinary Oxygenation (Amsterdam UMC only) | From end to start of surgery and from transfer to ICU until discharge or 48 hours postoperatively.
  Mean urinary partial oxygen pressure (PuO2)

CONTACTS AND LOCATIONS:
Overall Officials: Daniël H. van Raalte, MD, PhD, Principal Investigator — Internal Medicine Specialist
Locations (6):
- Netherlands (6):
  - OLVG, Amsterdam
  - Amsterdam UMC, Amsterdam
  - Amphia Hospital, Breda
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - St Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: Yes
Complete data collection methods and results will be shared with other researchers upon a formal request made to the principal investigator including a detailed motivation for the request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after peer-reviewed publication of the primary trail results.
Access Criteria: Official request made to the principal investigator.

REFERENCES:
- [Background] Semler MW, Rice TW, Shaw AD, Siew ED, Self WH, Kumar AB, Byrne DW, Ehrenfeld JM, Wanderer JP. Identification of Major Adverse Kidney Events Within the Electronic Health Record. J Med Syst. 2016 Jul;40(7):167. doi: 10.1007/s10916-016-0528-z. Epub 2016 May 27. PMID 27234478
- [Background] Myles PS, Shulman MA, Heritier S, Wallace S, McIlroy DR, McCluskey S, Sillar I, Forbes A. Validation of days at home as an outcome measure after surgery: a prospective cohort study in Australia. BMJ Open. 2017 Aug 18;7(8):e015828. doi: 10.1136/bmjopen-2017-015828. PMID 28821518
- [Background] Federici S, Bracalenti M, Meloni F, Luciano JV. World Health Organization disability assessment schedule 2.0: An international systematic review. Disabil Rehabil. 2017 Nov;39(23):2347-2380. doi: 10.1080/09638288.2016.1223177. Epub 2016 Nov 7. PMID 27820966
- [Background] Stolk E, Ludwig K, Rand K, van Hout B, Ramos-Goni JM. Overview, Update, and Lessons Learned From the International EQ-5D-5L Valuation Work: Version 2 of the EQ-5D-5L Valuation Protocol. Value Health. 2019 Jan;22(1):23-30. doi: 10.1016/j.jval.2018.05.010. Epub 2019 Jan 2. PMID 30661630
- [Background] Lau D, Pannu N, James MT, Hemmelgarn BR, Kieser TM, Meyer SR, Klarenbach S. Costs and consequences of acute kidney injury after cardiac surgery: A cohort study. J Thorac Cardiovasc Surg. 2021 Sep;162(3):880-887. doi: 10.1016/j.jtcvs.2020.01.101. Epub 2020 Mar 3. PMID 32299694
- [Background] Menne J, Dumann E, Haller H, Schmidt BMW. Acute kidney injury and adverse renal events in patients receiving SGLT2-inhibitors: A systematic review and meta-analysis. PLoS Med. 2019 Dec 9;16(12):e1002983. doi: 10.1371/journal.pmed.1002983. eCollection 2019 Dec. PMID 31815931
- [Background] Gilbert RE, Thorpe KE. Acute kidney injury with sodium-glucose co-transporter-2 inhibitors: A meta-analysis of cardiovascular outcome trials. Diabetes Obes Metab. 2019 Aug;21(8):1996-2000. doi: 10.1111/dom.13754. Epub 2019 May 24. PMID 31050116
- [Derived] Oosterom-Eijmael M, Monteiro de Oliveira NP, Niesten ED, Tolsma M, Snellen FT, Gerritse BM, Scohy TV, Rettig T, Godfried MB, Voogd MF, Wink J, van der Werff LM, Eberl S, Preckel B, Hermanides J, van Raalte DH, Hulst AH; MERCURI-2 study group. Study protocol of the multicentre, randomised, triple-blind, placebo-controlled MERCURI-2 trial: promoting effective renoprotection in cardiac surgery patients by inhibition of sodium glucose cotransporter (SGLT)-2. BMJ Open. 2025 May 16;15(5):e095504. doi: 10.1136/bmjopen-2024-095504. PMID 40379310